CLINICAL TRIAL: NCT07045870
Title: Effects of Perioperative Intravenous Lidocaine Infusion Versus Ketamine Infusion For Postoperative Analgesia in Patients Undergoing Thyroidectomy : A Randomized Controlled Trial
Brief Title: Methods of Post Operative Analgesia in Patients Undergoing Thyroidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mario Nashaat, Resident, Anasethesia, Surgical Icu, Pain management Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-6-11MS
Record Dates: First submitted 2025-06-21; First posted 2025-07-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Disorder
MeSH Terms: conditions — Thyroid Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- group L : will receive lidocaine (Active Comparator): lidocaine Infusion will be given for Postoperative Analgesia in Patients Undergoing Thyroidectomy
  Interventions: Drug: group L : will receive lidocaine
- group k : will receive ketamine (Active Comparator): Ketamine Infusion will be given for Postoperative Analgesia in Patients Undergoing Thyroidectomy
  Interventions: Drug: group k : will receive Ketamine
- group c: will receive .9% saline (Placebo Comparator): .9% saline will be given for Postoperative Analgesia in Patients Undergoing Thyroidectomy
  Interventions: Drug: group c: will recieve .9% saline

INTERVENTIONS:
Drug: group L : will receive lidocaine — group L : will receive 1.5 mg/kg bolus of iv lidocaine 10 minutes before anaesthesia induction then continuous iv infusion rate 1.5 mg / kg / h
  Arms: group L : will receive lidocaine
Drug: group k : will receive Ketamine — patients will receive .25 mg / kg bolus of iv ketamine 10 minutes before anaesthesia induction then continuous iv infusion of ketamine at .25 mg /kg /h
  Arms: group k : will receive ketamine
Drug: group c: will recieve .9% saline — group c will be injected with equivalent volumes and rates of .9% saline using the same application scheme as the lidocaine and ketamine as a control group
  Arms: group c: will receive .9% saline

SUMMARY:
this study aims to compare between effects of lidocaine and ketamine infusion on postoperative analgesia in patients undergoing thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 75 years old
* both sexes
* scheduled for thyroidectomy

Exclusion Criteria:

* toxic goiter
* (BMI) exceeding 30 kg / m2
* un controlled hypertension
* sever liver or kidney disorders
* allergy to study drugs
* hyperthyroidism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
the effect of perioperative intravenous lidocaine and ketamine infusion for postoperative analgesia in patients undergoing thyroidectomy | 24 hours posftoperative
  postoperative pain by Numerical Rating Scale (NRS) Zero means no pain and ten means worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Ludwig B, Ludwig M, Dziekiewicz A, Mikula A, Cisek J, Biernat S, Kaliszewski K. Modern Surgical Techniques of Thyroidectomy and Advances in the Prevention and Treatment of Perioperative Complications. Cancers (Basel). 2023 May 26;15(11):2931. doi: 10.3390/cancers15112931. PMID 37296896
- [Background] Javidi S, Sadrizadeh S, Sadrizadeh A, Bonakdaran S, Jarahi L. Postoperative complications and long-term outcomes after total and subtotal thyroidectomy: a retrospective study. Sci Rep. 2025 Jan 29;15(1):3705. doi: 10.1038/s41598-024-79860-8. PMID 39881145
- [Background] Jain SN, Lamture Y, Krishna M. Enhanced Recovery After Surgery: Exploring the Advances and Strategies. Cureus. 2023 Oct 17;15(10):e47237. doi: 10.7759/cureus.47237. eCollection 2023 Oct. PMID 38022245